CLINICAL TRIAL: NCT01737125
Title: Morphological Study of Distal Tibio-fibular Joint by Static MRI, Dynamics of Movement and Effort in Spatial High Resolution. Clinical Implication
Brief Title: Morphological Study of Distal Tibio-fibular Joint on MRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5318
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Distal Tibio-fibular Joint
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging (MRI) — * spatial high-resolution MRI multiplanar acquisition in T1 and T2 anatomical sequences
  * MRI acquisition in movements with dynamic sequences BEAT-IRT ( dynamic TrueFISP)

SUMMARY:
The distal tibio-fibular joint ( DTFJ) be an integral part of the ankle and its injury makes all the gravity, forecast and complexity of ankle fracture treatment. It's classically described and known by radiological point of view, but in static incidence and from anatomical studies. To our knowledge the dynamic dimension and its modelling is missing. Our study will use high spatial-resolution MRI acquisition to obtain the best possible definition of DTFJ but especially it will be associated with MRI acquisition in movement, using typical fast sequences " TrueFISP " and "FLASH" which will allow a precise modelling of joint physiological movements and biomechanics on healthy subjects by a not invasive method. This analysis will be made on a simple movement of flexion and extension, the other possible movements of the ankle being blocked what corresponds to the clinical situation of an osteosynthesis ankle immobilized in post-operative by a dynamic rehabilitation shoe Axmed ® It will be associated an"effort test " with the reproduction of subjected joint of a load with MRI joint movement control This test will be made with an ankle fixed to 90 ° of flexion what reproduces the post-operative clinical situationThe meditative data will be associated with an anatomical biomechanical study of ankles presenting a syndesmosis injury repaired according to the classic protocol using in our department, by comparing them with the data of the literature to optimize techniques repair of this joint. Indeed there is not gold standard surgical technique Main PurposeTo understand, observe, analyze and quantify the joint movement during a simple movement of ankle extension and flexion, and during a simulation of axial load miming walk fixed to 90 ° as in post-operative. Secondary purpose - Modelling the DTFJ- Modify the post-operative care with hypothesis that load does not lead abnormal movement in DTFJ with an ankle fixed to 90 ° ( post-operative clinical condition). - Validate our technique of repair of this joint by comparing the data MRI with anatomical mechanical tests

ELIGIBILITY:
Inclusion criteria:

* major subjects
* without ankle surgical antecedent
* Subject having signed an enlightened consent

Exclusion criteria:

* Subject in exclusion period
* Subject operated for the ankle,
* Impossibility to give an enlightened information
* Subject under protection of justice
* Under guardianship subject
* Patient refusing to participate in the study
* Minor subject
* Pregnant or breast-feeding woman
* Claustrophobic patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major subjects without ankle surgical antecedent
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu EHLINGER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Orthopédique et de Traumatologie, Hôpital de Hautepierre, Strasbourg, France